CLINICAL TRIAL: NCT04777682
Title: Intestinal Ultrasound Versus Double Balloon Enteroscopy (DBE) in Diagnosis of Malabsorption Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nada Abouelnaga Mahmoud, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: U.S V.S DBE in malabsorption
Record Dates: First submitted 2021-02-26; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Malabsorption Syndrome
MeSH Terms: conditions — Malabsorption Syndromes | interventions — High-Energy Shock Waves; Double-Balloon Enteroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Other): A single-arm, open, single-center (hospital-based) prospective interventional study to compare intestinal ultrasound versus double balloon enteroscopy in diagnosis of malabsorption syndrome
  Interventions: Procedure: ultrasound, double balloon enteroscopy

INTERVENTIONS:
Procedure: ultrasound, double balloon enteroscopy — compare intestinal ultrasound versus double-balloon enteroscopy in diagnosis of malabsorption syndrome

SUMMARY:
Our aim is to compare between intestinal ultrasound and double-balloon enteroscopy in the diagnosis of malabsorption syndrome.

DETAILED DESCRIPTION:
Malabsorption is impaired absorption of nutrients caused by any disruption in the process of normal absorption. Normal nutrient absorption requires 3 steps:

1. Luminal and brush border processing (e.g Celiac disease, crohn's disease, short bowel syndrome, radiation enteropathy, HIV enteropathy and drug-induced enteropathy).
2. Absorption into the intestinal mucosa.(e.g Lactose intolerance).
3. Transport into the circulation (e.g Primary intestinal lymphangiectasis, secondary obstructions from lymphoma, and infectious causes such as Whipple disease) (van der Heide, 2016).

Malabsorption may be either global or partial (isolated). Global malabsorption results from diseases with diffuse small bowel mucosal involvement or reduced absorptive surface, leading to impaired absorption of almost all nutrients (Keller and Layer, 2014).

Partial or isolated malabsorption results from diseases that interfere with the absorption of specific nutrients (van der Heide, 2016).

Malabsorption disorders are multifactorial, making diagnosis difficult. Symptoms are nonspecific and are frequently mistaken for other conditions, resulting in missed diagnoses . A comprehensive history can often be diagnostic. Several laboratory studies, imaging,and endoscopic evaluations are available to aid in diagnosing malabsorption disorders (Nikaki and Gupte ,2016).

The diagnosis of diseases involving the small bowel is challenging (black box of the gastrointestinal tract) due to the anatomy of this intestinal portion and the lack of tools for proper diagnosis (Jeon and Kim, 2013).

Despite recent advances in technology, endoscopic investigation of the small bowel remains challenging, with imaging techniques now playing an increasingly crucial role in the diagnosis and monitoring of diseases of the small bowel (Nylund et al.,2009).

Although computed tomography(CT)and fluoroscopic studies remain the gold standard investigations, both carry a significant radiation dose, so magnetic resonance imaging(MRI) and ultrasonography(US)are increasingly used as the first-line investigation, especially when imaging patients with inflammatory bowel disease where subsequent repeat imaging to monitor disease activity is useful, but the cumulative radiation dose from CT and fluoroscopic examinations is a concern (Panes et al., 2013).

Intestinal ultrasound has become an important diagnostic tool in the detection of bowel diseases. An advantage of ultrasound imaging compared with endoscopy and contrast radiography is that it permits evaluation of the transmural aspects of inflammatory or neoplastic pathology within its surrounding structures. Other advantages are that it is widely available, noninvasive, can be performed without preparation, and lacks radiation exposure (which may be particularly desirable in patients such as pregnant women) (Atkinson et al., 2017).

On the other hand, important limitations of ultrasonography are that the alimentary tract cannot be visualized over its entire length, many of the findings are nonspecific, and obtaining and interpreting the images is operator-dependent. Furthermore, ultrasound is far less useful in obese patients in whom high-frequency scanning may not be possible (Bryant et al., 2018).

There are three enteroscopy methods currently available: double balloon enteroscopy (DBE), single balloon enteroscopy and spiral enteroscopy. DBE was developed in 2001 by Hironori Yamamoto, and it began to be used in 2004. It enabled the visualization of almost all the bowel, DBE may be performed by anterograde or retrograde way, and the complete enteroscopy can be fulfilled by performing DBE by one extremity (Ferro et al., 2010).

The initial reason for the development of device assisted enteroscopy was the need for better endoscopic access to the small bowel in order to diagnose and/or treat intestinal pathology ( Ching et al.,2017).

Indications for DBE are multiple and are increasingly expanding because the procedure allows, besides the diagnosis of diseases, interventions like biopsies and other therapeutics ( Miranda 2014).

The most common indications for DBE are obscure gastrointestinal bleeding, Crohn's disease and celiac disease ( Ching et al.,2017).

The value of DBE for the surveillance and treatment of hereditary polyposis syndromes is clear ( Beggs et al.,2010).

Therapeutic options of DBE are diverse and comprehend any procedure performed during enteroscopy with diagnostic and curative purpose, including biopsy, polypectomy, argon plasma coagulation (APC), sclerotherapy with adrenaline injection and dilatation with balloon (Gurkan et al.,2013).

Other indications for DBE have since emerged. These new indications can be divided into the following categories: pediatric enteroscopy, DBE-assisted colonoscopy, (Tan et al.,2017) endoscopic access to gastrointestinal segments out of reach of conventional endoscopes and ERCP in patients with altered anatomy ( Cai et al.,2017).

Despite its long duration, DBE is a relatively safe procedure with a complication rate comparable to that of conventional endoscopic procedures ( L. Xin et al.,2011).

The most prevalent major complications are perforation, bleeding, acute pancreatitis and enteritis. Most commonly, there may be minor complications, which include abdominal discomfort and minimal trauma to the intestinal mucosa. It allows the patient to receive medical discharge in the same day ( Pata et al., 2010).

ELIGIBILITY:
Inclusion Criteria:

* Our study will include all patients referred to our unit with suspected malabsorption syndrome with one or more of the following will be included:

  1. Clinically:

     * Chronic watery, diurnal, and nocturnal, bulky, and frequent diarrhea.
     * Steatorrhea.
     * Abdominal pain and /or distention.
     * Anorexia, nausea, vomiting.
     * Weight loss.
     * Anemic manifestations
     * Vitamin deficiencies manifestations (e.g Bleeding, bruising, glossitis Peripheral neuropathy) Malnutrition and growth retardation in children.
     * Extraintestinal manifestations (e.g Dermatitis herpetiformis, Ankylosing spondylitis, erythema nodosum).
  2. Laboratory: routine blood tests that may reveal anemia, high CRP or low albumin, low calcium, and vitamin D level, high fecal calprotectin.

Exclusion Criteria:

* Mechanical gastrointestinal obstruction.
* Pregnant ladies.
* Those who fail to provide consent.
* Those unfit for anesthesia (with cardio-pulmonary embarrassment )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Intestinal Ultrasound Versus Double Balloon Enteroscopy (DBE) in Diagnosis of Malabsorption Syndrome | two years
  compare between intestinal ultrasound and double balloon enteroscopy in the diagnosis of malabsorption syndrome.

CONTACTS AND LOCATIONS:
Overall Officials: Laila Ab El-Touny, prof, Study Chair — Assuit University, Egypt; Khaled Ab Khalaf, Dr, Study Director — Assuit University, Egypt; Sayed Ha Ahmed, Dr, Study Director — Assuit University, Egypt; Nada A Mahmoud, Dr, Principal Investigator — Assuit University, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ching HL, McAlindon ME, Sidhu R. An update on small bowel endoscopy. Curr Opin Gastroenterol. 2017 May;33(3):181-188. doi: 10.1097/MOG.0000000000000346. PMID 28212152
- [Background] Ferro SM de, Correia JM, Pereira AD, Chavez P, Casaca R, Leitão CN. Divertículo de Meckel: diagnóstico por enteroscopia de duplo balão. 2010; 17: 65 - 8.
- [Background] Gurkan OE, Karakan T, Dogan I, Dalgic B, Unal S. Comparison of double balloon enteroscopy in adults and children. World J Gastroenterol. 2013 Aug 7;19(29):4726-31. doi: 10.3748/wjg.v19.i29.4726. PMID 23922469
- [Background] Jeon SR, Kim JO. Deep enteroscopy: which technique will survive? Clin Endosc. 2013 Sep;46(5):480-5. doi: 10.5946/ce.2013.46.5.480. Epub 2013 Sep 30. PMID 24143307
- [Background] Keller J, Layer P. The Pathophysiology of Malabsorption. Viszeralmedizin. 2014 Jun;30(3):150-4. doi: 10.1159/000364794. PMID 26288588
- [Background] Xin L, Liao Z, Jiang YP, Li ZS. Indications, detectability, positive findings, total enteroscopy, and complications of diagnostic double-balloon endoscopy: a systematic review of data over the first decade of use. Gastrointest Endosc. 2011 Sep;74(3):563-70. doi: 10.1016/j.gie.2011.03.1239. Epub 2011 May 28. PMID 21620401
- [Background] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Background] Nikaki K, Gupte GL. Assessment of intestinal malabsorption. Best Pract Res Clin Gastroenterol. 2016 Apr;30(2):225-35. doi: 10.1016/j.bpg.2016.03.003. Epub 2016 Mar 8. PMID 27086887
- [Background] Nylund K, Odegaard S, Hausken T, Folvik G, Lied GA, Viola I, Hauser H, Gilja OH. Sonography of the small intestine. World J Gastroenterol. 2009 Mar 21;15(11):1319-30. doi: 10.3748/wjg.15.1319. PMID 19294761
- [Background] Panes J, Bouhnik Y, Reinisch W, Stoker J, Taylor SA, Baumgart DC, Danese S, Halligan S, Marincek B, Matos C, Peyrin-Biroulet L, Rimola J, Rogler G, van Assche G, Ardizzone S, Ba-Ssalamah A, Bali MA, Bellini D, Biancone L, Castiglione F, Ehehalt R, Grassi R, Kucharzik T, Maccioni F, Maconi G, Magro F, Martin-Comin J, Morana G, Pendse D, Sebastian S, Signore A, Tolan D, Tielbeek JA, Weishaupt D, Wiarda B, Laghi A. Imaging techniques for assessment of inflammatory bowel disease: joint ECCO and ESGAR evidence-based consensus guidelines. J Crohns Colitis. 2013 Aug;7(7):556-85. doi: 10.1016/j.crohns.2013.02.020. Epub 2013 Apr 11. PMID 23583097
- [Background] Pata C, Akyuz U, Erzin Y, Mercan A. Double-balloon enteroscopy: the diagnosis and management of small bowel diseases. Turk J Gastroenterol. 2010 Dec;21(4):353-9. doi: 10.4318/tjg.2010.0120. PMID 21331987
- [Background] Prachayakul V, Deesomsak M, Aswakul P, Leelakusolvong S. The utility of single-balloon enteroscopy for the diagnosis and management of small bowel disorders according to their clinical manifestations: a retrospective review. BMC Gastroenterol. 2013 Jun 22;13:103. doi: 10.1186/1471-230X-13-103. PMID 23800178
- [Background] Tan M, Lahiff C, Bassett P, Bailey AA, East JE. Efficacy of Balloon Overtube-Assisted Colonoscopy in Patients With Incomplete or Previous Difficult Colonoscopies: A Meta-analysis. Clin Gastroenterol Hepatol. 2017 Oct;15(10):1628-1630. doi: 10.1016/j.cgh.2017.04.023. Epub 2017 Apr 19. No abstract available. PMID 28433783
- [Background] van der Heide F. Acquired causes of intestinal malabsorption. Best Pract Res Clin Gastroenterol. 2016 Apr;30(2):213-24. doi: 10.1016/j.bpg.2016.03.001. Epub 2016 Mar 8. PMID 27086886
- [Result] Atkinson NSS, Bryant RV, Dong Y, Maaser C, Kucharzik T, Maconi G, Asthana AK, Blaivas M, Goudie A, Gilja OH, Nuernberg D, Schreiber-Dietrich D, Dietrich CF. How to perform gastrointestinal ultrasound: Anatomy and normal findings. World J Gastroenterol. 2017 Oct 14;23(38):6931-6941. doi: 10.3748/wjg.v23.i38.6931. PMID 29097866
- [Result] Beggs AD, Latchford AR, Vasen HF, Moslein G, Alonso A, Aretz S, Bertario L, Blanco I, Bulow S, Burn J, Capella G, Colas C, Friedl W, Moller P, Hes FJ, Jarvinen H, Mecklin JP, Nagengast FM, Parc Y, Phillips RK, Hyer W, Ponz de Leon M, Renkonen-Sinisalo L, Sampson JR, Stormorken A, Tejpar S, Thomas HJ, Wijnen JT, Clark SK, Hodgson SV. Peutz-Jeghers syndrome: a systematic review and recommendations for management. Gut. 2010 Jul;59(7):975-86. doi: 10.1136/gut.2009.198499. PMID 20581245
- [Result] Bryant RV, Friedman AB, Wright EK, Taylor KM, Begun J, Maconi G, Maaser C, Novak KL, Kucharzik T, Atkinson NSS, Asthana A, Gibson PR. Gastrointestinal ultrasound in inflammatory bowel disease: an underused resource with potential paradigm-changing application. Gut. 2018 May;67(5):973-985. doi: 10.1136/gutjnl-2017-315655. Epub 2018 Feb 3. PMID 29437914
- [Result] Cai JX, Diehl DL, Kiesslich R, Storm AC, El Zein MH, Tieu AH, Hoffman A, Singh VK, Khashab MA, Okolo PI 3rd, Kumbhari V. A multicenter experience of through-the-scope balloon-assisted enteroscopy in surgically altered gastrointestinal anatomy. Surg Endosc. 2017 Jul;31(7):2753-2762. doi: 10.1007/s00464-016-5282-2. Epub 2016 Dec 30. PMID 28039647